CLINICAL TRIAL: NCT00456781
Title: GraftJacket® Rotator Cuff Tendon Reinforcement Scaffold: A Randomized Prospective Clinical Evaluation
Brief Title: Use of Graft Jacket for Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Collaborators: Sports Medicine & Arthroscopic Surgery Bone & Joint Clinic of Houston (Unknown); Southern California Orthopedic Institute Medical Group (Unknown); Kelsey-Seybold Clinic (Other); Plano Orthopedic & Sports Medicine Center (Unknown); St Joseph's Hospital Hand & Upper Limb Center (Unknown); Fowler Kennedy Sport Medicine Clinic (Other); St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Robert Litchfield, MD, FRCSC, Study Principal Investigator, Fowler Kennedy Sport Medicine Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wright1
Record Dates: First submitted 2007-02-21; First posted 2007-04-05 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Rotator Cuff Tear
Keywords: rotator cuff; randomized clinical trial
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augmentation (Experimental): Rotator Cuff Repair augmented with the Graft Jacket Device
  Interventions: Device: Augmentation
- No Augmentation (Active Comparator): Rotator Cuff RFepair
  Interventions: Device: Augmentation; Procedure: Rotator Cuff Repair without augmentation

INTERVENTIONS:
Device: Augmentation — Rotator Cuff Repair plus Graft Jacket
  Other Names: Wright Medical Technology Graft Jacket
Procedure: Rotator Cuff Repair without augmentation — Rotator Cuff Repair without augmentation
  Arms: No Augmentation

SUMMARY:
This study is to evaluate the safety and effectiveness of GraftJacket, a human tissue product used in fixing large and massive reparable rotator cuff tears.GraftJacket allograft (Wright Medical Technology, Inc., Arlington, TN) is a biologic tissue that is derived from human dermis. The primary purpose of this study is to determine whether rotator cuff repair augmentation using GraftJacket allograft provides a viable alternative, based on observed clinical outcomes, versus outcomes traditionally achieved with suture and anchor repairs. The study will secondarily investigate the difference in outcomes in patients treated arthroscopically versus open. This study will report patient progress and results at early (6 month) and late (2 year) time points in patients treated for large and massive reparable rotator cuff tears (>3cm). A reparable tear is defined as a tear of the rotator cuff where it is possible to bring the retracted tendon edge back to the greater tuberosity of the humerus without excessive tension. Restoration of rotator cuff integrity, clinical outcomes and re-tear rate will be included in the study evaluations.

DETAILED DESCRIPTION:
This is a prospective multi-center clinical study evaluating GraftJacket in the augmentation of large and massive rotator cuff tears compared to the traditional surgical technique of sutures and anchors alone. The study group will consist of 160 patients (early withdrawals or drop outs will not be replaced). Surgical approach for each patient will be either mini-open or arthroscopic. Safety assessments for this clinical study will be based on reported adverse events. Any adverse event that occurs during the study that represents a change from the patient's condition as noted at baseline [determined by normal standard of care] that is related to the procedure will be documented by completing the adverse events case report form.

Each investigator will indicate which operative technique (mini-open or arthroscopic) will be used during the study period at their site. The site selection process will be used to attempt to attain an equal distribution of both operative techniques used in the study. Patients will be randomly assigned to the treatment groups A or B. A randomization scheme using a 2 block model will be used within each surgical technique. Randomization cards meeting the requirements for this process will be generated by the statistician. Both surgical technique treatment groups will use the same assessments for comparisons throughout the study period.

Enrollment Plan for the GraftJacket Rotator Cuff Tendon Reinforcement Scaffold Surgical Technique Open Surgical (suture and anchor) Arthroscopic Group A without augmentation Group B with GraftJacket Group A without augmentation Group B with GraftJacket

Patients with reparable rotator cuff repairs must present with large and massive rotator cuff tears of more than 3cm, which can be repaired either arthroscopically or by open surgery to be eligible for enrollment. A reparable rotator cuff tear is defined as a tear of the rotator cuff where it is possible to bring the retracted tendon edge back to the greater tuberosity of the humerus without excessive tension. It should be possible to accomplish a watertight repair or only leave a residual defect of less than or equal to 1cm. The anteroposterior and mediolateral dimensions of the rotator cuff tear will be assessed intra-operatively by measurements either including the edges or after the edges are trimmed depending on the judgment of the surgeon. Rotator cuff tears involving the subscapularis tendon will not be included in the study, because the postoperative rehabilitation is more difficult and may confound the outcome results of either group. Surgical variables that should be documented on source documents and appropriate CRFs are the size of rotator cuff tear, the number of tendons involved, the type of repair (open, mini-open, arthroscopic) and the type and number of sutures and anchors.

Both clinical assessments and magnetic resonance imaging will be used to evaluate the effectiveness of the surgical techniques in both groups A and B. A screen/baseline MRI will be obtained of the affected shoulder during the preoperative visit. This MRI will be used to evaluate the extent of involvement and determine suitability for enrollment into the study including the size of the tear and extent of muscle atrophy. Images obtained within 3 months of signing consent may be used to assess eligibility for enrollment. Three additional follow-up MRIs of the affected shoulder will be obtained as part of the 2 year post-operative evaluation and will be used to evaluate structural success of group A, suture and anchor or group B, GraftJacket® allograft augmentation. The MRI scans performed at 6 months, 12 months and 24 months will be used to determine the rate of re-tear and to help to assess the integrity of the rotator cuff. Re-tears which are evident on the 6-month MRI will be considered a failure of the surgical technique, will be excluded from further follow-up within the study and followed separately. The comparison of the proportions of re-tears in patients in groups A and B who complete the MRI regimen through 2 years will be used to determine if GraftJacket® augmentation is a viable alternative to suture and anchor.

The Investigator will use clinical, functional, radiological, assessment of adverse events and assessment of the surgical techniques of groups A or B to evaluate each patient enrolled in this clinical study.

Pre Operative Procedures - Screen (Baseline)

Screening activities are performed during Visit 1. The protocol requires the following assessments during that visit:

* Informed consent process completed before any study related activities begin
* Inclusion/Exclusion criteria evaluation for study entry qualifications
* Magnetic Resonance Imaging (MRI)
* American Shoulder and Elbow Society (ASES) Scale
* University California Los Angeles (UCLA) Score
* Constant-Murley Score (CMS) Operative Procedures

The protocol requires completion of the following assessments during Visit 2:

* Open wound evaluation of rotator cuff tear for classification as large or massive with measurement of the tear to confirm size and length
* Enrollment confirmed using WMT randomization scheme for patient assignments Post Operative Procedures

Protocol requires the following assessments to be completed during the 1 month (plus 15 days) -Visit 3; 3 month (plus 15 days)-Visit 4; 6 month (plus 30 days) -Visit 5 and 12 month (plus 30 days) -Visit 6:

* MRI - Only performed during the 6 month (plus 30 day)-Visit 5 and 12 month (plus 30 days) -Visit 6
* ASES Scale
* CMS
* UCLA Score End of Study

Protocol requires completion of the following assessments during 24 month (plus 30 days)-Visit 7:

* MRI
* ASES Scale
* CMS
* UCLA Score
* Completion of End of Study Evaluation Form by the Principal Investigator

4.7 Scientific validity of the study design: Address the strengths and weaknesses of the selected design. Specifically indicate why a particular design was selected.

(1 page maximum - adhere to page limitations) Strengths: Prospective Randomized Clinical Trial Weakness: While not a true weakness, this trial is not randomized in the regular way but is using the "Expertise Randomization" style where the surgeon chooses his particular expertise of surgical repair of the rotator cuff (mini-open or arthroscopic) and the patients are randomized within that group.

A telephone randomization scheme cannot be used so there will be envelopes available to the surgeon in the OR for the group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18 - 75 years inclusive,
2. Reads, understand and able to complete the patient reported outcomes in English,
3. Patients with large and massive rotator cuff tears of more than 3cm, which can be repaired either arthroscopically or by open surgery.,
4. Patients with either primary or revision rotator cuff tears measuring < 5cm with at least 2 tendon involvement as indicated by MRI,
5. Patients who have a reasonable movement of the non-operative arm, defined as a shoulder elevation of equal or more than 90°, and are able to perform (postoperative) exercises,
6. Patients for whom there is a reasonable expectation that he or she will be available for each protocol required post-operative follow-up examination,
7. Patients must complete the informed consent process (including any regulatory requirements such as HIPAA authorization) agreeing to participate and signing the informed consent form prior to the site conducting any study related procedures.

Exclusion Criteria:

1. Patients with irreparable large or massive rotator cuff tears <3cm will be excluded if found intra-operatively
2. Patients with rotator cuff tears where the subscapularis tendon is disrupted,
3. Patients with inflammatory or auto-immune based joint diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus),
4. Patients with evidence of active infection, cancer, or highly communicable diseases that would preclude the patient from completing required patient assessments and clinic visits as described in the protocol,
5. Patients who smoke,
6. Patients with a documented history of drug abuse within six months of treatment,
7. Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment.
8. Females of child-bearing potential who are pregnant or breastfeeding, or plan to become pregnant during the course of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
less or no recurrence of shoulder rotator cuff tear with the use of the tissue scaffold than with the standard use of surgical anchors and screws as measured by MRI results | 2 years
  each subject will be eligible for the study based on the Pre-operative results of the MRI as it relates to the size of the tissue tear. The subjects will be assigned to either the tissue scaffold material or the standard surgical suture or anchors. Then, the procedure to repair is determined by the investigator as an arthoscopic or open procedure. Pos-operative evalutions via MRI will be obtained throughout the study to evaluate the effectiveness of the surgical procedure and for the measurement of retear or not.

SECONDARY OUTCOMES:
Scale (pain, ADL, Shoulder stability) | 2 years
  A baseline evaluation for pain scale, activity of daily living measurement and range of motion to determine injured and repaired shoulder stability
UCLA Shoulder Score (pain, function, manual muscle testing) | 2 years
  Pain, function, manual muscle testing measured per UCLA Shoulder Score at baseline and at intervals at up to two years.
Constant-Murley Shoulder Score (pain, function, ROM, Strength) | 2 years
  Pain, function, ROM, and Strength measured per Constant-Murley Shoulder Score at baseline and at intervals at up to two years.
Surgeon Reported Satisfaction | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Litchfield, MD, FRCSC, Principal Investigator — Fowler Kennedy Sport Medicine Clinic
Locations (7):
- United States (4):
  - Southern California Orthopedic Institute, Simi Valley, California
  - Bone and Joint Clinic of Houston, Houston, Texas
  - Kelsey-Seybold Orthopedic, Houston, Texas
  - Plano Orthopedic & Sports Medicine, Plano, Texas
- Canada (3):
  - Pan Am Clinic, Winnipeg, Manitoba
  - Fowler Kennedy Sport Medicine Clinic, London, Ontario
  - The Hand and Upper Limb Centre, London, Ontario